CLINICAL TRIAL: NCT03668249
Title: Characterization of a Multidimensional Model to Predict the Course of Crohn's Disease: A Pilot Study
Brief Title: A Study to Characterize Multidimensional Model to Predict the Course of Crohn's Disease (CD)
Acronym: PREMONITION-CD
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: IBD-5002; U1111-1220-0873 (Registry Identifier: WHO)
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease
Keywords: Drug therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants diagnosed with CD from approximately 12 to 15 investigational sites will be observed retrospectively for previous 5 years.

SUMMARY:
The descriptive purpose of this study is to characterize clinical and nonclinical factors of participants with CD, participant flow and visits to other specialists in the hospitals of the healthcare network of the Autonomous Community of Madrid with implementation of electronic medical records. The clinical and nonclinical factors include: demographic and baseline clinical characteristics, lifestyle, relapses, complications, day hospital visits, surgery, presence of complications such as perianal fistulas and complex perianal fistulas. The predictive purpose of this study is to develop a statistical predictive model with the information obtained from the descriptive purpose, in the hospitals of the healthcare network of the Autonomous Community of Madrid, capable of assigning any participant diagnosed with CD a probability of reaching a prototypical clinical condition or a probability of experiencing certain clinical complications.

DETAILED DESCRIPTION:
This is a retrospective and non-interventional study of participants with CD. The study will collect data from electronic medical records (EMRs) of the participants in the hospitals of the healthcare network of the Autonomous Community of Madrid with implementation of EMRs and will describe the determining factors and develop a statistical model for predicting likely outcomes in participants with CD. This study will conduct an additional substudy to evaluate the performance of the system through a human assessment to be performed by the clinical experts at each participating site.

The study will have a retrospective data collection from EMRs of the participants referring to last 5 years.

The study will enroll approximately 3000 participants. All participants will be enrolled in one observational cohort.

This multi-center trial will be conducted in Spain. The overall time for data collection in the study will be approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with CD from the medical centers participating in the study.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants diagnosed with CD, will be observed retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 5938 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants who had Relapses | Approximately 5 years
Number of Participants who had Disease Related Complications | Approximately 5 years
Number of day Hospital Visits | Approximately 5 years
Number of Participants who had Surgeries | Approximately 5 years
Number of Participants with Complications Such as Perianal Fistulas and Complex Perianal Fistulas | approximately 5 years
Participant Flow | Approximately 5 years
Number of Participants who Visit to Other Specialists | Approximately 5 years

SECONDARY OUTCOMES:
Prevalence of the Different Phenotypes | Approximately 5 years
  Development of a statistical predictive model capable of assigning any patient diagnosed with CD a probability of reaching a prototypical clinical condition or a probability of experiencing certain clinical complications.
Number of Participants who met the Eligibility Criteria to Receive Biological Treatment for CD | Approximately 5 years
Number of Direct and Indirect Resources Used | Approximately 5 years
  Health care resources of participants with CD will be assessed in terms of direct and indirect resources. Direct resources will include number of hospital admissions, emergency and hospital visits, and tests performed, etc. Indirect resources related to decreased productivity of CD participants through a specific variable, the total number of work days lost due to CD during the study period.
Number of Essential Factors on Which Physician's Predictions of Participant Outcomes are Based | Approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (8):
- Spain (8):
  - HM Hospitales, Boadilla, Madrid
  - H. U. de Fuenlabrada, Fuenlabrada, Madrid
  - H.U. Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - H.U. Rey Juan Carlos, Móstoles, Madrid
  - H.U. Infanta Sofia, San Sebastián de los Reyes, Madrid
  - H. U. Infanta Elena, Valdemoro, Madrid
  - H Infanta Leonor y Virgen de la Torre, Vallecas, Madrid
  - H La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Gomollon F, Gisbert JP, Guerra I, Plaza R, Pajares Villarroya R, Moreno Almazan L, Lopez Martin MC, Dominguez Antonaya M, Vera Mendoza MI, Aparicio J, Martinez V, Tagarro I, Fernandez-Nistal A, Lumbreras S, Mate C, Montoto C; Premonition-CD Study Group. Clinical characteristics and prognostic factors for Crohn's disease relapses using natural language processing and machine learning: a pilot study. Eur J Gastroenterol Hepatol. 2022 Apr 1;34(4):389-397. doi: 10.1097/MEG.0000000000002317. PMID 34882644